CLINICAL TRIAL: NCT06496724
Title: A Clinical Study of Albumin-bound Paclitaxel/Granulocyte-based Therapy for Recurrent/Metastatic Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: JIANG LONGWEI (Other)
Collaborators: China Pharmaceutical University (Unknown)
Responsible Party: Sponsor-Investigator, JIANG LONGWEI, associate researcher, Jinling Hospital, China
Organization: Jinling Hospital, China (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: swzl20230906
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Albumin paclitaxel/neutrophil drug (Experimental): Isolate the patients' autologous neutriphil cells, induce and culture them with albumin paclitaxel in vitro. Then the drug will be infused intravenously into patients. The number of neutriphil cells will be more than 1.0E10.
  Interventions: Biological: Albumin paclitaxel/neutrophil drug

INTERVENTIONS:
Biological: Albumin paclitaxel/neutrophil drug — Isolate the patients' autologous neutriphil cells, induce and culture them with albumin paclitaxel in vitro. The final product for Albumin paclitaxel/neutrophil drug.

SUMMARY:
The goal of this clinical trial is to learn if Albumin-bound Paclitaxel/Granulocyte drug can treat patients with recurrent/metastatic breast cancer. The main questions it aims to answer are:

To verify the safety of Albumin-bound Paclitaxel/Granulocyte drug in patients with recurrent/metastatic breast cancer.

To evaluate the efficacy of Albumin-bound Paclitaxel/Granulocyte drug in patients with recurrent/metastatic breast cancer.

To detect the pharmacokinetic behavior of Albumin-bound Paclitaxel/Granulocyte drug in patients with recurrent/metastatic breast cancer.

DETAILED DESCRIPTION:
In this open, single-armed study, selected patients with recurrent/metastatic breast cancer confirmed by Histopathology will be received Albumin-bound Paclitaxel/Granulocyte-based therapy. The granulocyte will be separated by blood cell separator, and will be cultured in the GMP laboratory to make Albumin-bound Paclitaxel/Granulocyte drug. Then the drug will be infused intravenous into patients.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged ≥ 18 years old; Obtain an informed consent form voluntarily signed by the patient themselves; Recurrent/metastatic advanced breast cancer patients (refer to TNM standard); Patients who have received standard first-line treatments and expected survival time ≥ 3 months; EOCG score ≤ 2 and KPS≥ 70 points; Liver, kidney and bone marrow functions are basically normal; Patients of childbearing age need to take appropriate protective measures before enrollment and after treatment 3 months.

Exclusion Criteria:

* Individuals who have received other anti-tumor treatment within 4 weeks prior the enrollment; Patients with history of allergy to paclitaxel, albumin naproxen, ibuprofen, trimethoprim and ampicillin; Positive blood pregnancy test; Patients who required anti coagulant therapy; Patients with active infectious diseases or a history of bone marrow or organ transplantation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
To verity the safety of Albumin-bound Paclitaxel/Granulocyte in the treatment of Recurrent/Metastatic Breast Cancer | 13 months
  The adverse events and severe adverse events will be evaluated.

SECONDARY OUTCOMES:
To evaluate the efficiency of Albumin-bound Paclitaxel/Granulocyte drug in the treatment of Recurrent/Metastatic Breast Cancer | 13 months
  The objective clinical response will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Jia Shaochang, MD, Study Director — Jinling Hospital, China
Locations (1):
- Jinling Hospital, Nanjing, Jiangsu, China